CLINICAL TRIAL: NCT05125939
Title: Improving Colonoscopy Adenoma Detection Metrics by Extending the Screening-only Measurement to All Indications: a Prospective Multicenter Study
Brief Title: Can Overall Adenoma Detection Rate Replace Screening Adenoma Detection Rate ? Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Evergreen General Hospital, Taiwan (Other)
Collaborators: E-DA Hospital (Other); E-Da Dachang Hospital (Unknown); Chang Gung Memorial Hospital (Other); Sepulveda Ambulatory Care Center, Veterans Affairs Greater Los Angeles Healthcare System (Unknown)
Responsible Party: Sponsor
Other Study IDs: EGH-2022-1
Record Dates: First submitted 2021-11-07; First posted 2021-11-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Adenoma Detection Rate; Colonoscopy
Keywords: Colonoscopy; Adenoma detection rate; Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Screening indication: Screening indication includes asymptomatic patients aged ≥50 years with no prior colonoscopy and at average risk of CRC. Screening indication also includes asymptomatic patients with negative prior colonoscopy.
  Interventions: Other: Comparison of ADR
- Surveillance indication: Surveillance indication includes patients with prior colon neoplasms, including conventional adenomas and clinically significant serrated polyps.
  Interventions: Other: Comparison of ADR
- Diagnostic indication: Diagnostic indication includes patients who report symptoms (e.g., abdominal pain, a change in bowel habits, or rectal bleeding) before their first screening examination and undergo evaluation of an abnormality on other image study, unexplained anemia and/or unexplained weight loss.
  Interventions: Other: Comparison of ADR
- Positive fecal immunochemical test: FIT+ indication includes patients who undergo colonoscopy for positive FIT results in screen-eligible individuals. FIT+ indication also applies to those with a positive FIT result and a recent colonoscopy.
  Interventions: Other: Comparison of ADR

INTERVENTIONS:
Other: Comparison of ADR — The investigators will compare ADRs using traditional screening-restricted definition and combined screening, surveillance, and diagnostic indication (i.e., overall-non-FIT indication). The impact of addition of FIT+ indication into the overall indication (i.e., overall-FIT indication) on ADR will also be evaluated.

SUMMARY:
This is a prospective equivalence colonoscopy study evaluating whether overall adenoma detection rate (ADR) is a reliable alternate for screening ADR. Overall indication includes screening, surveillance, and diagnostic indications.

DETAILED DESCRIPTION:
This multicenter study will be conducted by 18 colonoscopists from 5 hospitals in Taiwan, including Evergreen general hospital, E-da hospital, E-da Dachang hospital, Linkou Chang Gung memorial hospital, and Keelung Chang Gung memorial hospital, and plans to recruit 2700 prospective participants in a 2-year period. Felix W. Leung from Sepulveda Ambulatory Care Center, Veterans Affairs Greater Los Angeles Healthcare System (USA) will be involved in the study design, and will participate in data analyses and report preparation. Consecutive patients aged ≥50 years undergoing colonoscopy are eligible for enrollment. Positive fecal immunochemical test (FIT+) is considered as an independent indication category and the colonoscopy indications are categorized into 4 groups: screening, surveillance, diagnostic, and FIT+. Overall indication will be subdivided into overall excluding FIT (overall-non-FIT) group and overall including FIT (overall-FIT) group. In this study, the investigators plan to (1) compare individual ADR across 4 colonoscopy indication categories (screening, surveillance, diagnostic, FIT+); (2) explore correlations between screening ADR and overall-non-FIT and overall-FIT ADRs, respectively.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients aged ≥50 years undergoing colonoscopy are eligible for enrollment.

Exclusion Criteria:

* high risk family history of colorectal cancer (CRC) e.g., familial adenomatous polyposis, hereditary non-polyposis CRC syndrome, multiple first degree relatives with CRC, or a single first degree relative with CRC at <60 years
* serrated polyposis syndrome
* inflammatory bowel disease
* colonoscopy to remove a large neoplastic polyps
* obstructive lesions of the colon
* gastrointestinal bleeding
* current participation in other studies
* hospitalized patients
* mental retardation
* pregnancy
* refusal to provide a written informed consent.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥50 years undergoing screening, surveillance, diagnostic, and FIT+ colonoscopy are eligible for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 7 days
  The proportion of participants undergoing a complete colonoscopy who have one or more adenomas detected

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Liang Cheng, Principal Investigator — Evergreen General Hospital, Taoyuan, Taiwan
Locations (6):
- Sepulveda Ambulatory Care Center, VAGLAHS, North Hills, California, United States
- Taiwan (5):
  - E-Da Dachang Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - Evergreen General Hospital, Taoyuan District
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kahi CJ, Vemulapalli KC, Johnson CS, Rex DK. Improving measurement of the adenoma detection rate and adenoma per colonoscopy quality metric: the Indiana University experience. Gastrointest Endosc. 2014 Mar;79(3):448-54. doi: 10.1016/j.gie.2013.10.013. Epub 2013 Nov 15. PMID 24246797
- [Background] Kaltenbach T, Gawron A, Meyer CS, Gupta S, Shergill A, Dominitz JA, Soetikno RM, Nguyen-Vu T, A Whooley M, Kahi CJ. Adenoma Detection Rate (ADR) Irrespective of Indication Is Comparable to Screening ADR: Implications for Quality Monitoring. Clin Gastroenterol Hepatol. 2021 Sep;19(9):1883-1889.e1. doi: 10.1016/j.cgh.2021.02.028. Epub 2021 Feb 19. PMID 33618027
- [Background] Rex DK, Ponugoti PL. Calculating the adenoma detection rate in screening colonoscopies only: Is it necessary? Can it be gamed? Endoscopy. 2017 Nov;49(11):1069-1074. doi: 10.1055/s-0043-113445. Epub 2017 Jul 28. PMID 28753699
- [Background] Ladabaum U, Shepard J, Mannalithara A. Adenoma and Serrated Lesion Detection by Colonoscopy Indication: The ADR-ESS (ADR Extended to all Screening/Surveillance) Score. Clin Gastroenterol Hepatol. 2021 Sep;19(9):1873-1882. doi: 10.1016/j.cgh.2021.04.027. Epub 2021 Apr 22. PMID 33895358